CLINICAL TRIAL: NCT03585530
Title: Raltitrexed Concurrent With Radiotherapy for Elderly Chinese Patients With Squamous Cell Carcinoma of Esophagus: A Phase-II Study
Brief Title: Raltitrexed Concurrent With Radiotherapy for Elderly Chinese Patients With Squamous Cell Carcinoma of Esophagus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Huai'an First People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: huaianzhuweiguo1
Record Dates: First submitted 2018-07-01; First posted 2018-07-13 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Esophagus Squamous Cell Carcinoma
Keywords: Esophageal neoplasma; adjuvant therapy; raltitrexed; radiotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — raltitrexed

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental)
  Interventions: Drug: raltitrexed

INTERVENTIONS:
Drug: raltitrexed — Raltitrexed 2.6mg/m2 was administered on d1、d22

SUMMARY:
Concurrent chemoradiotherapy is one of the curative options for esophageal squamous cell carcinoma. We evaluated the efficacy and toxicity of raltitrexed with concurrent radiotherapy in elderly patients with esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

Histological or cytologic diagnosis of esophageal carcinoma. ECOG performance status 0-1. Age:70-85 years. Joined the study voluntarily and signed informed consent form Patients must not have received any prior anticancer therapy.

Stage IIa-Ⅳa(AJCC 2002). Target lesions can be measured according to RECIST criteria. No serious system dysfunction and immuno-deficiency, Adequate organ function including the following: Hemoglobin ≥9 g/dL, WBC≥3x109/L, Neutrophils (ANC )≥1.5x109/L, platelet count ≥100x 109/L, TBIL<1.5 x ULN, ALT and AST ≦ 2.5 x ULN, creatinine ≦ 1.5 x ULN.

Exclusion Criteria:

Multiple carcinomas of the esophagus. Biopsy-proven invasion of the tracheobronchial tree or tracheoesophageal fistula.

Metastatic disease (M1b). A primary tumor that extended to within 2 cm of the gastroesophageal junction. Prior chemotherapy, prior thoracic radiation, surgical resection of the primary tumor.

history of a second malignancy other than nonmelanoma skin cancer.

Ages: 70 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-03-15 (Estimated)

PRIMARY OUTCOMES:
Overall survival(OS) | 3 years
  From the date of randomization until the date of death

SECONDARY OUTCOMES:
Disease-free survival (DFS) | 3 years
  From the date of randomization to the date of first observation of disease progression, or relapse, or death due to any cause
treatment-related toxicities | From the date of randomization until six months after treatment completion
  Toxicities were graded according to the National Cancer Institute Common Toxicity Criteria (NCICTC), version 3.0
Quality of life(QOL) | 3 years
  QOL is respectively evaluated at randomization and 1 month, 3 month, 6 month and yearly after treatment among patients by using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C-30 (EORTC QLQ-C30)

CONTACTS AND LOCATIONS:
Locations (1):
- Huai'an First Hospital, Huai'an, Jiangsu, China